CLINICAL TRIAL: NCT03032198
Title: "Early R&D Clinical Evaluation of Opto-Acoustic Tomography for Detection and Diagnostic Differentiation of Thyroid Nodules"
Brief Title: "Clinical Evaluation of Opto-Acoustic Tomography for Detection and Diagnostic Differentiation of Thyroid Nodules"
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Revision to over all corporate strategy
Sponsor: Seno Medical Instruments Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Thyroid-01
Record Dates: First submitted 2017-01-20; First posted 2017-01-26 (Estimated); Results first posted 2022-07-13 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-07

CONDITIONS: Feasibility Study for Thyroid Indication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Imagio OA/US Scan (Experimental): Imagio opto-acoustic gray-scale ultrasound scan
  Interventions: Device: Imagio OA/US

INTERVENTIONS:
Device: Imagio OA/US — Diagnostic opto-acoustic gray-scale ultrasound
  Other Names: opto-acoustic gray-scale ultrasound

SUMMARY:
Thyroid Feasibility Study

DETAILED DESCRIPTION:
This is an early R&D Feasibility study to assess Imagio OA/US's ability to optimize the device algorithm specific to thyroid in order to detect the difference between benign and malignant thyroid nodules

ELIGIBILITY:
Inclusion Criteria:

1. Have been informed of the nature of the study and provided written informed consent, prior to initiation of any study activities;
2. Have an undiagnosed suspicious solid or mostly solid thyroid nodule.;
3. 18 years of age or older at the time of consent;
4. Are willing and able to complete all procedures and assessments in accordance with the clinical protocol; and,
5. Have received recommendation for and are scheduled for an ultrasound guided FNAB, ultrasound guided core biopsy, excisional biopsy, lobectomy or complete thyroidectomy of at least one thyroid nodule.

Exclusion Criteria:

1. Are prisoners;
2. Have a condition or impediment (i.e., insect bites, poison ivy, open sores, chafing of the skin, scar, tattoos, moles, etc.); that could interfere with the intended field of view (within one probe length or 4 cm of the nodule),
3. Previous or on-going radioactive iodine treatment.
4. Nodule to be biopsied is greater than 3.0 cm in maximum diameter;
5. Is pregnant;
6. Have an acute or a chronic hematoma and/or acute ecchymosis of the thyroid;
7. Is experiencing photo-toxicity or photo-sensitivity or is undergoing treatment for a photo-sensitive condition such as porphyria or lupus erythematosus;
8. Patient has received chemotherapy for any type of cancer within 90 days from date of screening CDU;
9. Have had previous image guided FNAB or surgical biopsy of the target nodule of interest within the 45 days of baseline Imagio Scan;
10. Patient has participated in a clinical study of an investigational drug or device within 3 months prior to screening CDU that may have an impact on clinical outcomes; and,
11. Patient has previously participated in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2017-12-04 (Actual); Primary Completion 2018-06-17 (Actual); Study Completion 2019-04-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tom Stavros, MD, Principal Investigator — Seno Medical, Inc.
Locations (2):
- United States (2):
  - Invision Sally Jobe, Greenwood Village, Colorado
  - UT Health Science Center, San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Trial was terminated early due to corporate strategy changes
Period: Overall Study
Arm/Group | Imagio OA/US Scan
Started | 37
Completed (Trial was terminated early due to change in corporate strategy) | 36
Not Completed | 1
Not completed — Screen Fail | 1

BASELINE CHARACTERISTICS:
Population: 36 patients under-going an Imagio exam, 1 screen failure prior to Imagio exam
Arm/Group | Imagio OA/US Scan
Number analyzed (Participants) | 37
Age, Continuous [Median (Standard Deviation); unit: Years] | 57 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 32
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 36
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 37

OUTCOME MEASURES:

1. Primary Outcome: Initial Assessment of Imagio's Ability to Distinguish Between Benign and Malignant Thyroid Nodules.
Description: The primary objective of this feasibility study is to provide an initial assessment of Imagio OA's ability to distinguish between benign and malignant thyroid nodules, and when appropriate, between benign and metastatic cervical lymph nodes in subjects.
Time Frame: 12-24 months
Population: This Early R&D Development Study was terminated early due to change in corporate strategy. The study was discontinued before we initiated the independent reader portion of the study which would have been the basis for producing the data that is needed for analyzing this endpoint.
Arm/Group | Imagio OA/US Scan
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: AEs were collected during Imagio scanning at baseline
Arm/Group | Imagio OA/US Scan
All-Cause Mortality (participants affected / at risk) | 1/36
Serious Adverse Events (participants affected / at risk) | 0/36
Other Adverse Events (participants affected / at risk) | 1/36
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Imagio OA/US Scan (N=36)
Pain (General disorders) | 1 (1) — One subject reported pain due to pressure of the OA probe related to the depth of lesion. This event was brief and resolved without treatment

LIMITATIONS AND CAVEATS:
The study was discontinued due to change in corporate strategy. This Early R&D Development Study was terminated early due to change in corporate strategy. The reader portion of the study was not initiated per the protocol, therefore was no data generated for the primary and secondary endpoints to analyze.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-06): https://cdn.clinicaltrials.gov/large-docs/98/NCT03032198/Prot_SAP_000.pdf